CLINICAL TRIAL: NCT04521205
Title: A Multicenter Clinical Trial: Efficacy, Safety of Fecal Microbiota Transplantation for Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMZSYY-AF-SC-12-03
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Disease, Ulcerative Colitis Type
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized FMT (Experimental): The patients will receive standardized FMT. The FMT was given by capsule. It was given three times a week.
  Interventions: Drug: fecal microbiota capsule
- Without FMT (Placebo Comparator): The patients will receive FMT with blank capsule.
  Interventions: Drug: fecal microbiota capsule

INTERVENTIONS:
Drug: fecal microbiota capsule — a capsule full of fecal microbiota extracting from the health

SUMMARY:
There are many limitations in the current treatments of Inflammatory bowel disease(IBD). Some patients have no or little reaction to the traditional drugs. Now the investigators realized that the intestinal microbiota is closely associated with the development of IBD. In recent years, a retrospective study showed that the overall efficiency of fecal microbiota transplantation (FMT) for IBD was 79%, the overall remission rate was 43%, which opened a new chapter in the treatment of IBD. So the standardized fecal microbiota transplantation is considered to be simple but effective emerging therapies for the treatment of IBD. In this project the investigators intend to carry out a single-center, randomized, single-blind clinical intervention study. The investigators plan to recruit patients with IBD (Ulcerative Colitis and Crohn's Disease) in China. The patients will be randomly divided into two groups, one group will be given treatment of standardized fecal microbiota transplantation, the other will be simply treated with traditional drugs, followed up for at least 1 year. The investigators aim to determine the efficiency, durability and safety of Fecal Microbiota Transplantation for IBD treatment, and further to explore which major microbiota may effect in this project.

DETAILED DESCRIPTION:
In this projects the investigators aim to re-establish a gut balance of intestinal microbiota through Standardized Fecal Microbiota Transplantation for IBD (UC and CD). We have established a standardized isolation, store, and transport steps of fecal bacteria from donated fresh stool in the laboratory. Then the bacteria will be transplanted to mid-gut by capsule. Patients in this study will be assigned to receive standardized FMT three times or not and would be followed up for at least 1 year. The clinical symptoms, sign, blood tests, endoscopy and questionnaire will be used to assess the efficiency, durability and safety of Standardized FMT at the start and end of the projects. At last, we will use 16S-rDNA to estimate the change of intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Standard or conventional medicine treatment ineffective of IBD patients
2. IBD patients with recurrent symptoms
3. IBD patients who had drug dependence or recurrence when reduced or discontinued use
4. Untreated IBD patients who voluntarily received FMT

Exclusion Criteria:

1. IBD patients with contraindications for gastrointestinal endoscopy
2. IBD patients combined with other serious diseases such as respiratory failure, heart failure and severe immunodeficiency
3. IBD patients with indication of surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission: the modified Mayo score and endoscopy | up to one year
  Clinical remission defined as modified Mayo score≦2 (range 0-12). The endpoint of follow-up is the time of clinical recurrence. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanyun Fan, Xiamen, China

IPD SHARING:
Plan to Share IPD: No